CLINICAL TRIAL: NCT02129244
Title: A Nurse Case Management Intervention to Improve MDR-TB/HIV Co-Infection Outcomes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Medical Research Council, South Africa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NA_00078899; RO1 104488-01A1 (Other Grant/Funding Number: NIH/NAID)
Record Dates: First submitted 2014-04-29; First posted 2014-05-02 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: MDR-TB; HIV
Keywords: MDR-TB; HIV; Nurse Case Management (NCM)
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NCM Plus Intervention (Active Comparator): The researchers designed the NCM-Plus intervention by integrating the domains of the Chronic Care Model with added attention to linkage to care, building on evidence-based guidelines and the team's pilot findings. In the NCM bundle, the researchers provide extensive details on both proximal and distal outcome variables. Nurse case managers will be hired and trained to improve disease management for patients with MDR-TB and HIV. Specific measurable responsibilities will be implemented by each NCM at sites randomized to receive the intervention. The NCM-patient interaction will occur at the MDR-TB treatment inpatient or outpatient facility.
  Interventions: Other: NCM-Plus
- Standard/Usual Care (No Intervention): Usual care is defined as standardized programmatic management of MDR-TB/HIV without care coordination. Nurses are present as part of the team, but with no special coordination role, leaving the MDR-TB physician solely responsible for treatment outcomes with little support. Physicians see patients weekly during the intensive phase and the patient receives basic daily nursing care without coordination of care, active monitoring of Adverse Drug Reactions (ADR)s or HIV care integration. This care transitions to monthly visits with the physician in the continuation phase, again with very little nursing involvement in care coordination.

INTERVENTIONS:
Other: NCM-Plus — The NCM will follow the domains of the chronic care model by:
  1. Assuring effective, efficient clinical care and self-management support
  2. Promoting clinical care consistent with scientific evidence and patient preferences
  3. Organizing data to facilitate efficient, effective care
  4. Empowering and preparing patients to manage their health and health-care needs
  5. Mobilizing community resources to meet the needs of patients
  Arms: NCM Plus Intervention

SUMMARY:
The researchers of this study are observing the treatment of multi-drug resistant Mycobacterium tuberculosis (MDR-TB) in South Africa. MDR-TB can not be treated with the usual TB drugs and needs to be treated with special drugs. The patients need to take these drugs for up to two years. Certain hospitals have already agreed to participate in this research project, half of the hospitals will be assigned a nurse case manager and the other half will not. The researchers are studying the benefits of having a nurse case manager to improve treatment response for patients with drug resistant TB. The researchers believe that nurse case management (NCM) in the intervention sites will increase MDR-TB cure and completion rates (i.e. treatment success) in comparison to usual care (UC), i.e. standardized programmatic management alone, in patients with and without HIV co-infection. To do this, the researchers will review the medical information collected at the hospital as part of the patient's treatment after obtaining the patient's permission.

DETAILED DESCRIPTION:
Mycobacterium tuberculosis (TB) remains the leading cause of death among persons living with Human Immunodeficiency Virus/Acquired Immunodeficiency Syndrome (HIV/AIDS) in southern Africa. This syndemic places an overwhelming burden on healthcare workers and the health system. Drug-resistant TB remains a growing threat to public health despite advances in treatment and diagnosis over the past decade. South Africa has the world's highest rate of TB/HIV co-infection and ranks fourth worldwide for both multi-drug resistant (MDR) TB incidence and HIV prevalence. Treatment of MDR-TB, defined as resistance to isoniazid and rifampin, remains challenging and its treatment course complex. Success of second line treatment regimens is considerably less likely than first line treatment with significantly more adverse drug reactions (ADRs). Prospective cohort studies from South Africa report less than 50% treatment success (i.e. cure or completion) and significant differences in patients with and without HIV are noted. Differences in sex and gender as well as age are rarely evaluated. In addition to the management complexity and length of treatment, systems level factors such as access to care and healthcare capacity contribute to poorer treatment outcomes. Insufficient numbers of trained physicians capable and clinically competent to manage the challenges of integrated MDR-TB/HIV care are commonplace. These circumstances place a heavy burden on the most abundant healthcare resource in South Africa, the nurse. Nurses with proficiency in care models for both diseases are essential to improve treatment outcomes. The investigators experience dictates, however, that patients endure lengthy treatment with little assessment, support or guidance from nursing professionals due to a lack of training as well as lack of evidence-based interventions and delineated models of care for MDR-TB patients.

Nurse case management (NCM) models in which a registered nurse facilitates and coordinates treatment plans to ensure that timely, evidence-based care is given improves treatment outcomes. Presently, there is little evidence to describe such models in TB/HIV co-infected patients globally, and specifically less evidence for MDR-TB/HIV in sub-Saharan Africa. Many studies, however, have demonstrated substantial improvements in disease outcomes utilizing nurse case managers. Complex diseases such as heart failure, diabetes, HIV and drug susceptible TB are among these. Substantial gaps remain, however, in the investigators understanding of the impact of such interventions among co-infected patients, the influence of such models among different age groups or the cost-benefit in under resourced settings. Prior studies provide strong evidence that interventions must be multi-faceted and foster system level approaches to improve treatment outcomes (i.e. NCM patient-centered care services coupled with systems level approaches to care coordination). The Chronic Care Model identifies essential elements of a health care system that encourage high-quality chronic disease care in such a systems approach. These elements provide the conceptual model and implementation structure for the proposed NCM plus health systems strengthening (i.e. NCM-plus) intervention, a multi-faceted health systems and patient-centered intervention to improve MDR-TB/HIV treatment outcomes. The proposed 5-year cluster randomized trial, will evaluate the NCM-plus intervention on MDR-TB treatment outcomes in South Africa, the epicenter of the MDR-TB/HIV epidemic.

Primary Aim:

To determine the impact of a NCM model (i.e. NCM-Plus) on MDR-TB outcomes in patients with and without HIV co-infection in South Africa through a cluster randomized trial.

Hypothesis:

Nurse case management (NCM) in intervention sites will increase MDR-TB cure and completion rates (i.e. treatment success) in comparison to usual care (UC), i.e. standardized programmatic management alone, in patients with and without HIV co-infection.

Secondary Aims:

1. To conduct sub-group analysis by a) HIV co-infection; b) sex and gender; and c) age
2. To compare the frequency and time to identification of adverse drug events between intervention and control sites.
3. To conduct a costing analysis and a cost-effectiveness evaluation of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Center (Cluster Level)

  1. MDR-TB Centers in KwaZulu-Natal (KZN) or Eastern Cape (EC), South Africa providing standardized
  2. MDR-TB regimen according to National Department of Health guidelines
  3. Facility has provided MDR-TB care for a minimum of 6 months at study initiation
  4. MDR-TB Centers with facility-based access to anti-retroviral therapy
  5. Facility willingness to participate in the study
* Individual (Patient Level)

  1. Patients 18 years of age and older, with microbiologically confirmed MDR- TB, admitted to receive inpatient care at a participating hospital who signs informed consent within 7 days of admission.
  2. Patients 13 - 17 years of age, with microbiologically confirmed MDR- TB, who provide consent for study team to contact parent or legal guardian and when patient is willing and parent or legal guardian provides approval for study participation within 7 days of admission.

Exclusion Criteria (Individual Patient Level):

* Persons who present to the MDR-TB ward who have started MDR-TB treatment prior to admission.
* Children, less than 13 years of age; only one participating center has an MDR-TB wards for children under 13.
* Persons who are unable or unwilling to provide informed consent for participation
* Any patient enrolled in another clinical trial that changes standard MDR- TB or HIV care.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3600 (Estimated)
Dates: Start 2014-10 (Actual); Primary Completion 2021-03 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who experience successful treatment outcomes | 24-36 months
  General Estimating Equations (GEE) Regression Analysis

SECONDARY OUTCOMES:
Proportion of patients who experience successful treatment outcomes based on HIV co-infection | 24 to 36 months
  Multivariate Analysis using binomial or Poisson-based GEE models
Proportion of patients who experience successful treatment outcomes based on sex and gender | 24-36 months
  Multivariate Analysis using binomial or Poisson-based GEE models
Proportion of patients who experience successful treatment outcomes based on age | 24-36 months
  Multivariate Analysis using binomial or Poisson-based GEE models

CONTACTS AND LOCATIONS:
Overall Officials: Jason E Farley, PhD, MPH, NP, Principal Investigator — Johns Hopkins University
Locations (15):
- South Africa (15):
  - Regus Primary Office, Westville, Durban
  - Catherine Booth Hospital, aMatikulu, KwaZulu-Natal
  - Don McKenzie, Durban
  - King George V Hospital, Durban
  - Fort Gray Hospital, East London
  - Dunstan Farrell Hospital, Hibberdene
  - Hlabisa Hospital, Hlabisa
  - Manguzi, Manguzi
  - Nkqubela, Mdantsane
  - Fosa Hospital, Newlands West
  - Doris Goodwin Hospital, Pietermaritzburg
  - Marjorie Parrish Hospital, Port Alfred
  - Jose Pearson Hospital, Port Elizabeth
  - Murchison Hospital, Port Shepstone
  - St Margaret's MDR-TB Hopsital, Umzimkulu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] World Health Organization. Global Tuberculosis Control. WHO/HTM/TB/2010.7. 2010. Geneva, Switzerland.
- [Background] World Health Organization. Multidrug and extensively drug-resistant TB (M/XDR-TB): 2010 global report on surveillance and response. [WHO/HTM/TB/2010.3]. 2010. World Health Organization, 20 Avenue Appia, 1211 Geneva 27, Switzerland, WHO Press.
- [Background] Orenstein EW, Basu S, Shah NS, Andrews JR, Friedland GH, Moll AP, Gandhi NR, Galvani AP. Treatment outcomes among patients with multidrug-resistant tuberculosis: systematic review and meta-analysis. Lancet Infect Dis. 2009 Mar;9(3):153-61. doi: 10.1016/S1473-3099(09)70041-6. PMID 19246019
- [Background] Johnston JC, Shahidi NC, Sadatsafavi M, Fitzgerald JM. Treatment outcomes of multidrug-resistant tuberculosis: a systematic review and meta-analysis. PLoS One. 2009 Sep 9;4(9):e6914. doi: 10.1371/journal.pone.0006914. PMID 19742330
- [Background] Farley JE, Ram M, Pan W, Waldman S, Cassell GH, Chaisson RE, Weyer K, Lancaster J, Van der Walt M. Outcomes of multi-drug resistant tuberculosis (MDR-TB) among a cohort of South African patients with high HIV prevalence. PLoS One. 2011;6(7):e20436. doi: 10.1371/journal.pone.0020436. Epub 2011 Jul 22. PMID 21799728
- [Background] Shean KP, Willcox PA, Siwendu SN, Laserson KF, Gross L, Kammerer S, Wells CD, Holtz TH. Treatment outcome and follow-up of multidrug-resistant tuberculosis patients, West Coast/Winelands, South Africa, 1992-2002. Int J Tuberc Lung Dis. 2008 Oct;12(10):1182-9. PMID 18812049
- [Background] Gandhi NR, Shah NS, Andrews JR, Vella V, Moll AP, Scott M, Weissman D, Marra C, Lalloo UG, Friedland GH; Tugela Ferry Care and Research (TF CARES) Collaboration. HIV coinfection in multidrug- and extensively drug-resistant tuberculosis results in high early mortality. Am J Respir Crit Care Med. 2010 Jan 1;181(1):80-6. doi: 10.1164/rccm.200907-0989OC. Epub 2009 Oct 15. PMID 19833824
- [Background] Somma D, Thomas BE, Karim F, Kemp J, Arias N, Auer C, Gosoniu GD, Abouihia A, Weiss MG. Gender and socio-cultural determinants of TB-related stigma in Bangladesh, India, Malawi and Colombia. Int J Tuberc Lung Dis. 2008 Jul;12(7):856-66. PMID 18544216
- [Background] O'Donnell MR, Zelnick J, Werner L, Master I, Loveday M, Horsburgh CR, Padayatchi N. Extensively drug-resistant tuberculosis in women, KwaZulu-Natal, South Africa. Emerg Infect Dis. 2011 Oct;17(10):1942-5. doi: 10.3201/eid1710.110105. PMID 22000378
- [Background] Vella V, Racalbuto V, Guerra R, Marra C, Moll A, Mhlanga Z, Maluleke M, Mhlope H, Margot B, Friedland G, Shah NS, Gandhi NR. Household contact investigation of multidrug-resistant and extensively drug-resistant tuberculosis in a high HIV prevalence setting. Int J Tuberc Lung Dis. 2011 Sep;15(9):1170-5, i. doi: 10.5588/ijtld.10.0781. PMID 21943840
- [Background] National Department of Health, South Africa. Decentralized Management of Multi-Drug Resistant Tuberculosis: A Policy Framework for South Africa. 2011.
- [Background] Welch G, Garb J, Zagarins S, Lendel I, Gabbay RA. Nurse diabetes case management interventions and blood glucose control: results of a meta-analysis. Diabetes Res Clin Pract. 2010 Apr;88(1):1-6. doi: 10.1016/j.diabres.2009.12.026. Epub 2010 Feb 8. PMID 20116879
- [Background] Nyamathi A, Nahid P, Berg J, Burrage J, Christiani A, Aqtash S, Morisky D, Leake B. Efficacy of nurse case-managed intervention for latent tuberculosis among homeless subsamples. Nurs Res. 2008 Jan-Feb;57(1):33-9. doi: 10.1097/01.NNR.0000280660.26879.38. PMID 18091290
- [Background] Del Sindaco D, Pulignano G, Minardi G, Apostoli A, Guerrieri L, Rotoloni M, Petri G, Fabrizi L, Caroselli A, Venusti R, Chiantera A, Giulivi A, Giovannini E, Leggio F. Two-year outcome of a prospective, controlled study of a disease management programme for elderly patients with heart failure. J Cardiovasc Med (Hagerstown). 2007 May;8(5):324-9. doi: 10.2459/JCM.0b013e32801164cb. PMID 17443097
- [Background] Anaya HD, Hoang T, Golden JF, Goetz MB, Gifford A, Bowman C, Osborn T, Owens DK, Sanders GD, Asch SM. Improving HIV screening and receipt of results by nurse-initiated streamlined counseling and rapid testing. J Gen Intern Med. 2008 Jun;23(6):800-7. doi: 10.1007/s11606-008-0617-x. Epub 2008 Apr 18. PMID 18421508
- [Background] Andersen MD, Smereck GA, Hockman EM, Ross DJ, Ground KJ. Nurses decrease barriers to health care by "hyperlinking" multiple-diagnosed women living with HIV/AIDS into care. J Assoc Nurses AIDS Care. 1999 Mar-Apr;10(2):55-65. doi: 10.1016/S1055-3290(06)60299-9. PMID 10065410
- [Background] Schumann A, Nyamathi A, Stein JA. HIV risk reduction in a nurse case-managed TB and HIV intervention among homeless adults. J Health Psychol. 2007 Sep;12(5):833-43. doi: 10.1177/1359105307080618. PMID 17855466
- [Background] Nyamathi AM, Christiani A, Nahid P, Gregerson P, Leake B. A randomized controlled trial of two treatment programs for homeless adults with latent tuberculosis infection. Int J Tuberc Lung Dis. 2006 Jul;10(7):775-82. PMID 16848340
- [Background] Hsieh CJ, Lin LC, Kuo BI, Chiang CH, Su WJ, Shih JF. Exploring the efficacy of a case management model using DOTS in the adherence of patients with pulmonary tuberculosis. J Clin Nurs. 2008 Apr;17(7):869-75. doi: 10.1111/j.1365-2702.2006.01924.x. PMID 17850292
- [Background] Wagner EH, Glasgow RE, Davis C, Bonomi AE, Provost L, McCulloch D, Carver P, Sixta C. Quality improvement in chronic illness care: a collaborative approach. Jt Comm J Qual Improv. 2001 Feb;27(2):63-80. doi: 10.1016/s1070-3241(01)27007-2. PMID 11221012
- [Background] Wagner EH, Bennett SM, Austin BT, Greene SM, Schaefer JK, Vonkorff M. Finding common ground: patient-centeredness and evidence-based chronic illness care. J Altern Complement Med. 2005;11 Suppl 1:S7-15. doi: 10.1089/acm.2005.11.s-7. PMID 16332190
- [Background] Institute of Medicine (US) Committee on Envisioning a Strategy for the Long-Term Burden of HIV/AIDS: African Needs and U.S. Interests. Preparing for the Future of HIV/AIDS in Africa: A Shared Responsibility. Washington (DC): National Academies Press (US); 2011. Available from http://www.ncbi.nlm.nih.gov/books/NBK209740/ PMID 24983048
- [Background] Joint United Nations Programme on HIV/AIDS (UNAIDS). Global Report: UNAIDS Report on the Global AIDS Epidemic, 2010. UNAIDS/10.11E | JC1958E. 2010.
- [Background] National Department of Health, South Africa. Decentalized Management of Multi-Drug Resistant Tuberculosis: A Policy Framework for South Africa. 2010.
- [Background] Department of Labour. The shortage of Medical Doctors in South Africa: Scarce and critical skills research project. 1-30-2009.
- [Background] National Department of Health, South Africa. Programmatic Management of Multi-Drug Resistant Tuberculosis: Emergency Update. 2008.
- [Background] Laserson KF, Thorpe LE, Leimane V, Weyer K, Mitnick CD, Riekstina V, Zarovska E, Rich ML, Fraser HS, Alarcon E, Cegielski JP, Grzemska M, Gupta R, Espinal M. Speaking the same language: treatment outcome definitions for multidrug-resistant tuberculosis. Int J Tuberc Lung Dis. 2005 Jun;9(6):640-5. PMID 15971391
- [Background] Brust JC, Gandhi NR, Carrara H, Osburn G, Padayatchi N. High treatment failure and default rates for patients with multidrug-resistant tuberculosis in KwaZulu-Natal, South Africa, 2000-2003. Int J Tuberc Lung Dis. 2010 Apr;14(4):413-9. PMID 20202298
- [Background] Lin RL, Lin FJ, Wu CL, Peng MJ, Chen PJ, Kuo HT. Effect of a hospital-based case management approach on treatment outcome of patients with tuberculosis. J Formos Med Assoc. 2006 Aug;105(8):636-44. doi: 10.1016/S0929-6646(09)60162-5. PMID 16935764
- [Background] Nathanson E, Nunn P, Uplekar M, Floyd K, Jaramillo E, Lonnroth K, Weil D, Raviglione M. MDR tuberculosis--critical steps for prevention and control. N Engl J Med. 2010 Sep 9;363(11):1050-8. doi: 10.1056/NEJMra0908076. No abstract available. PMID 20825317
- [Background] Department of Health. Management of Drug Resistant Tuberculosis: Policy Guidelines. i-151. 8-1-2012.
- [Background] Department of Health. National Strategic Plan on HIV, STIs and TB (2012-2016). 1-78. 12-1-2012.
- [Background] Boulle A, Clayden P, Cohen K, Cohen T, Conradie F, Dong K, Geffen N, Grimwood A, Hurtado R, Kenyon C, Lawn S, Maartens G, Meintjes G, Mendelson M, Murray M, Rangaka M, Sanne I, Spencer D, Taljaard J, Variava E, Venter WD, Wilson D. Prolonged deferral of antiretroviral therapy in the SAPIT trial: did we need a clinical trial to tell us that this would increase mortality? S Afr Med J. 2010 Sep 7;100(9):566, 568, 570-1. doi: 10.7196/samj.4434. No abstract available. PMID 20822639
- [Background] Dheda K, Lampe FC, Johnson MA, Lipman MC. Outcome of HIV-associated tuberculosis in the era of highly active antiretroviral therapy. J Infect Dis. 2004 Nov 1;190(9):1670-6. doi: 10.1086/424676. Epub 2004 Sep 29. PMID 15478074
- [Background] National Department of Health, South Africa. The South African Antiretroviral Treatement Guidelines 2010. 2010. 2010.
- [Background] Iseman MD. Treatment and implications of multidrug-resistant tuberculosis for the 21st century. Chemotherapy. 1999;45 Suppl 2:34-40. doi: 10.1159/000048480. PMID 10449896
- [Background] Weyer K, Brand J, Lancaster J, Levin J, van der Walt M. Determinants of multidrug-resistant tuberculosis in South Africa: results from a national survey. S Afr Med J. 2007 Nov;97(11 Pt 3):1120-8. No abstract available. PMID 18250922
- [Background] Amuha MG, Kutyabami P, Kitutu FE, Odoi-Adome R, Kalyango JN. Non-adherence to anti-TB drugs among TB/HIV co-infected patients in Mbarara Hospital Uganda: prevalence and associated factors. Afr Health Sci. 2009 Aug 1;9 Suppl 1(Suppl 1):S8-15. PMID 20589161
- [Background] Swaminathan S, Narendran G, Venkatesan P, Iliayas S, Santhanakrishnan R, Menon PA, Padmapriyadarsini C, Ramachandran R, Chinnaiyan P, Suhadev M, Sakthivel R, Narayanan PR. Efficacy of a 6-month versus 9-month intermittent treatment regimen in HIV-infected patients with tuberculosis: a randomized clinical trial. Am J Respir Crit Care Med. 2010 Apr 1;181(7):743-51. doi: 10.1164/rccm.200903-0439OC. Epub 2009 Dec 3. PMID 19965813
- [Background] Cramm JM, Finkenflugel HJ, Moller V, Nieboer AP. TB treatment initiation and adherence in a South African community influenced more by perceptions than by knowledge of tuberculosis. BMC Public Health. 2010 Feb 17;10:72. doi: 10.1186/1471-2458-10-72. PMID 20163702
- [Background] Kliiman K, Altraja A. Predictors and mortality associated with treatment default in pulmonary tuberculosis. Int J Tuberc Lung Dis. 2010 Apr;14(4):454-63. PMID 20202304
- [Background] Holtz TH, Lancaster J, Laserson KF, Wells CD, Thorpe L, Weyer K. Risk factors associated with default from multidrug-resistant tuberculosis treatment, South Africa, 1999-2001. Int J Tuberc Lung Dis. 2006 Jun;10(6):649-55. PMID 16776452
- [Background] Gardam M, Verma G, Campbell A, Wang J, Khan K. Impact of the patient-provider relationship on the survival of foreign born outpatients with tuberculosis. J Immigr Minor Health. 2009 Dec;11(6):437-45. doi: 10.1007/s10903-008-9221-8. Epub 2009 Jan 6. PMID 19127431
- [Background] Bloss E, Kuksa L, Holtz TH, Riekstina V, Skripconoka V, Kammerer S, Leimane V. Adverse events related to multidrug-resistant tuberculosis treatment, Latvia, 2000-2004. Int J Tuberc Lung Dis. 2010 Mar;14(3):275-81. PMID 20132617
- [Background] National Department of Health, South Africa. Decentralized Management of Multi-Drug Resistant Tuberculosis: A Policy Framework for South Africa (Draft). 2010.
- [Background] Guidelines for the Programmatic Management of Drug-Resistant Tuberculosis: 2011 Update. Geneva: World Health Organization; 2011. Available from http://www.ncbi.nlm.nih.gov/books/NBK148644/ PMID 23844450
- [Background] Wagner EH, Austin BT, Davis C, Hindmarsh M, Schaefer J, Bonomi A. Improving chronic illness care: translating evidence into action. Health Aff (Millwood). 2001 Nov-Dec;20(6):64-78. doi: 10.1377/hlthaff.20.6.64. PMID 11816692
- [Background] Moulton LH. Covariate-based constrained randomization of group-randomized trials. Clin Trials. 2004;1(3):297-305. doi: 10.1191/1740774504cn024oa. PMID 16279255
- [Background] Institute of Healthcare Improvement. Improving HIV Care: A Modular Quality Improvement Curriculum. Institue of Healthcare Improvemnet . 6-15-2011.
- [Background] Farley JE, Alwood K, Davis JG, Stellenberg E, and van der Walt M. Development and Pilot Testing of MDR-TB/HIV In-Service Training in Rural KwaZulu Natal. National Education Association and Foundation of Nursing University Deans of South Africa Annual Conference . 10-15-2010.
- [Background] Farley JE, Tudor C, Mphahlele M, Franz K, Perrin NA, Dorman S, Van der Walt M. A national infection control evaluation of drug-resistant tuberculosis hospitals in South Africa. Int J Tuberc Lung Dis. 2012 Jan;16(1):82-9. doi: 10.5588/ijtld.10.0791. PMID 22236851
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Roberts C, Roberts SA. Design and analysis of clinical trials with clustering effects due to treatment. Clin Trials. 2005;2(2):152-62. doi: 10.1191/1740774505cn076oa. PMID 16279137
- [Background] Campbell MK, Fayers PM, Grimshaw JM. Determinants of the intracluster correlation coefficient in cluster randomized trials: the case of implementation research. Clin Trials. 2005;2(2):99-107. doi: 10.1191/1740774505cn071oa. PMID 16279131
- [Background] Campbell MK, Mollison J, Grimshaw JM. Cluster trials in implementation research: estimation of intracluster correlation coefficients and sample size. Stat Med. 2001 Feb 15;20(3):391-9. doi: 10.1002/1097-0258(20010215)20:33.0.co;2-z. PMID 11180309
- [Background] Zeger SL, Liang KY. Longitudinal data analysis for discrete and continuous outcomes. Biometrics. 1986 Mar;42(1):121-30. PMID 3719049
- [Background] Gallop R, Small DS, Lin JY, Elliott MR, Joffe M, Ten Have TR. Mediation analysis with principal stratification. Stat Med. 2009 Mar 30;28(7):1108-30. doi: 10.1002/sim.3533. PMID 19184975
- [Background] Dumas JE, Lynch AM, Laughlin JE, Phillips Smith E, Prinz RJ. Promoting intervention fidelity. Conceptual issues, methods, and preliminary results from the EARLY ALLIANCE prevention trial. Am J Prev Med. 2001 Jan;20(1 Suppl):38-47. doi: 10.1016/s0749-3797(00)00272-5. PMID 11146259
- [Derived] McNabb KC, Bergman AJ, Patil A, Lowensen K, Mthimkhulu N, Budhathoki C, Perrin N, Farley JE. Travel distance to rifampicin-resistant tuberculosis treatment and its impact on loss to follow-up: the importance of continued RR-TB treatment decentralization in South Africa. BMC Public Health. 2024 Feb 23;24(1):578. doi: 10.1186/s12889-024-17924-0. PMID 38389038